CLINICAL TRIAL: NCT02352181
Title: Management of Coagulopathy During Orthotopic Liver Transplantation. Comparison Between ROTEM-based Management and Standard Biological Assessment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-870
Record Dates: First submitted 2014-12-18; First posted 2015-02-02 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplantation
Keywords: Cirrhosis, transplantation, transfusion, Rotem®
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S group (Placebo Comparator): S Group: will be transfused patients according to standard management based on conventional coagulation profile of the laboratory
  Interventions: Procedure: Conventional coagulation profile Analysis
- R group (Experimental): The R group will consist of patients transfused according to an algorithm based on the data of the coagulation ROTEM analysis.
  Interventions: Procedure: Rotem analysis

INTERVENTIONS:
Procedure: Conventional coagulation profile Analysis — Transfusional protocol for Standard group Red Blood cells concentrate if Hemoglobin <9 gram per liter Fibrinogen 3 gram, if fibrinogen <1gram per liter
  Platelet concentrate :
  * if platelets <50gram per liter before transfusion, at anhepatic phase, or in case of bleeding.
  * if platelets <30gram per liter at vascular unclamping time at the end of intervention or without bleeding 2 Fresh frozen plasma if :
  * if prothrombin<40% before transfusion at anhepatic phase or in case of bleeding.
  * if prothrombin<30% at vascular unclamping time at the end of intervention or without bleeding Bolus Tranexamic acid 1g and 3g every 24 hours in case of fibrin degradation products.
  Analyses common to both groups: NFS, chemistry panel with ionized serum calcium, blood gas with lactates, HemoCue ®, capillary blood glucose.
  Analyses in S Group only: coagulation profile (PT, APTT, INR, fibrinogen, platelet count, soluble complexes, PDF).
  Arms: S group
Procedure: Rotem analysis — Transfusional protocol for Rotem group. Red Blood cells concentrate if Hemoglobin <9 gram per liter Fibrinogen 3 gram, if A10 FIBTEM <8 mm
  Platelet concentrate :
  * If MCF EXTEM <40mm or A10<35 mm and MCF or A10 FIBTEM >8mm.
  * If platelets <30gram per liter at vascular unclamping time at the end of intervention or without bleeding.
    2 Fresh frozen plasma if CT EXTEM >100s.
  Bolus Tranexamic acid 1g and 3g every 24 hours :
  * if fibrinolysis in EXTEM
  * Reduction of 15 % of clotting time or clot formation time and increase of maximum clot firmness in APTEM compared to EXTEM, or maximal lysis at 60 minutes >15%.
  Analyses in R group only: blood sampling on citrated tube for ROTEM analysis (EXTEM, INTEM, FIBTEM, APTEM +/- HEPTEM), coagulation profile (same as that of the S Group, for emergency procedure).
  Analyses common to both groups: NFS, chemistry panel with ionized serum calcium, blood gas with lactates, HemoCue ®, capillary blood glucose.
  Arms: R group

SUMMARY:
In current practice, management of coagulation during liver transplantation is performed either through standard coagulation status or with ROTEM® depending on practitioner choice and availability of materials. In this context, the ROTEM® is used since over 2 years by anesthesiologists in the digestive surgery department of the Croix Rousse hospital in Lyon, France.

Indeed liver transplantation surgery is at high risk of bleeding due to coagulopathy developed by patients who are eligible, due to coagulation factor synthesis deficiencies in the cirrhotic liver. On the other hand the standard coagulation profile is a poor reflection of coagulopathy in such patients because the imbalance between pro- and anti-coagulant factors are not taken into account by PT and aPTT measures. Management of intraoperative hemorrhage may be facilitated by the ROTEM® which is performed from whole blood and which allows the detection of abnormalities in the balance between pro- and anti-coagulant factors.

This technique was already evaluated in liver, cardiac, and obstetric surgery but also in traumatology. Randomized trials in liver transplantation surgery have shown changes in transfusion practices but did not focus on the consequences of such changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients >=18 years of age
* Patients undergoing orthotopic liver transplantation in the Croix-Rousse Hospital within 24 months after inclusion and who have received clear information and who are not opposed to the participation in the study
* Patients affiliated to a social security system or similar
* Patients not subject to a measure of legal protection

Exclusion Criteria:

* Opposition to participation in the study
* Patients <18 years of age
* Patients who participated in the previous month to another study protocol
* Pregnant women or breast-feeding
* Not affiliated to a social security system
* Patients with hemostasis pathology (hemophilia, ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Amount of blood product (in milliliter) transfused during liver transplantation. | During time of liver transplantation an average of 9 hours.
  Assessing the impact of intraoperative management of coagulation by ROTEM® compared to the conventional management (standard coagulation profile) on the amount of blood product units (in milliliter) transfused during liver transplantation.

SECONDARY OUTCOMES:
Occurrence of serious respiratory complication. | within 48 first hours after liver transplantation.
  reintubation; acute pulmonary oedema.
Occurrence of thrombotic complication. | within 48 first hours after liver transplantation.
  hepatic artery thrombosis, sus hepatic thrombotic, portal thrombosis.
Occurrence of serious infectious complication | within 48 first hours after liver transplantation.
  septic shock; serious sepsis, intubation necessity for sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Bonnet, PH, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Bonnet A, Gilquin N, Steer N, Gazon M, Quattrone D, Pradat P, Maynard M, Mabrut JY, Aubrun F. The use of a thromboelastometry-based algorithm reduces the need for blood product transfusion during orthotopic liver transplantation: A randomised controlled study. Eur J Anaesthesiol. 2019 Nov;36(11):825-833. doi: 10.1097/EJA.0000000000001084. PMID 31567574